CLINICAL TRIAL: NCT00981240
Title: A Dose Escalation Safety and Pharmacokinetic Study of SAR103168 Administered as a Single Agent by Intravenous Infusion, Once Daily for 5 Consecutive Days to Patients With Refractory/ Relapsed Acute Leukemias or High-risk Myelodysplastic Syndromes.
Brief Title: Dose Escalation, Safety and Pharmacokinetic Study of SAR103168 in Patients Refractory/ Relapsed Acute Leukemias or High-risk Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED10416
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Acute Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — SAR103168

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose escalation (Experimental): Cohorts of 3 to 6 patients will be included at each dose level. The starting dose is 1.2mg/m2/day. The dose will be increased in new cohorts of patients according to toxicities observed during the first 4-week treatment period. The escalation process will continue until the MTD is determined. Additional 15 patients will be included at the MTD.
  Interventions: Drug: SAR103168

INTERVENTIONS:
Drug: SAR103168 — Pharmaceutical form: Concentrate for solution for infusion
  Route of administration: Intravenous infusion

SUMMARY:
Primary objectives:

* To determine the maximum tolerated dose (MTD) of SAR103168 and to characterize the dose limiting toxicities (DLTs) in the proposed dose regimen
* To evaluate the pharmacokinetic (PK) profile of SAR103168

Secondary objectives:

* To characterize the global safety profile of SAR103168
* To evaluate preliminary anti-leukemia activity
* To investigate the potential induction effect on CYP3A4 and persistence of this effect by using oral midazolam as a probe substrate in patients enrolled into the expanded cohort at the MTD
* To determine the metabolic pathways of SAR103168 and identify the chemical structures of metabolites
* To determine the potential impact of SAR103168 on the QTc interval in patients enrolled at the MTD

DETAILED DESCRIPTION:
Patients will receive the study drug until unacceptable toxicity, clinically significant disease progression, withdrawal of consent or investigator's decision, and for a maximum of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory/relapsed acute leukemias or high-risk myelodysplastic syndromes with no curative option available including any of the following:

  * Patients with de novo or secondary acute myelogenous leukemia (AML) (except acute promyelocytic leukemia), meeting one of the following conditions:
  * Refractory or relapsed AML; In case of first relapse the CR duration should be less than 12 months. If the relapse failed at least one prior salvage attempt, the CR duration may be more than 12 months.
  * Into the expanded cohort at the MTD, previously untreated AML patients over age 60 with poor- risk cytogenetics who are not eligible for or do not accept induction chemotherapy may also be included.
* Patients with refractory/relapsed acute lymphoblastic leukemia (ALL)
* Patients with high-risk myelodysplastic syndrome (MDS) as defined by the International Prognostic Scoring System
* Patients with chronic myeloid leukemia in blast phase (CML-BP)

Exclusion Criteria:

* performance status > 2
* Active uncontrolled central nervous system leukemia
* Cytotoxic therapy within 2 weeks prior to the first dose of SAR103168. For the non cytotoxic agents/investigational drugs this washout period should be at least 2 weeks or at least 5 half-lives whichever is longer. Hydroxyurea must be stopped at least 24 hours prior to the first dose of SAR103168
* Lack of recovery from toxicities from prior therapies to grade < 1
* White blood cells > 30 x 10^9/L prior to the first dose of SAR103168
* Prior allogeneic stem cell transplantation or donor lymphocytes infusion within 3 months preceding the first dose of SAR103168
* Any of the following within 6 months prior to the first dose of SAR103168:

  * Myocardial infarction, congestive heart failure, documented angina pectoris, arrhythmia requiring medication (in particular atrial fibrillation or flutter), severe conduction disorder (second or third atrio-ventricular block, pacemaker), coronary/peripheral artery bypass graft surgery
  * Arterial or venous thromboembolism, deep venous thrombosis
* Left ventricular ejection fraction < 50% by echocardiography or multiple gated acquisition scan
* Cardiac ischemia on 12-lead ECG
* Baseline QTc-interval > 500 msec
* Hypertension uncontrolled with appropriate therapy
* Active infection (viral, bacterial or fungal) uncontrolled with appropriate therapy
* Major surgery within 6 weeks prior to the first dose of SAR103168
* Poor organ function defined by one of the following:

  * Total bilirubin > 1.5 x upper limit of normal (ULN) unless related to leukemia (i.e. hemolysis) or Gilbert's syndrome
  * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 2.5 x ULN
  * Serum creatinine > 1.5 x ULN or calculated creatinine clearance < 50 mL/min
* Patients under treatment with potent inhibitors of CYP3A4 unless these treatments may be stopped at least 3 days prior to the first dose of SAR103168
* Patients under treatment with CYP3A4 or CYP2C9 inducers, unless these treatments may be stopped at least 3 days prior to the first dose of SAR103168
* Pregnant or breast-feeding women or refusal to use adequate contraceptive method, when applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Incidence of DLTs during the initial 4-week period of treatment | 4 weeks
Pharmacokinetic parameters of SAR103168 | First course: Days 1, 2, 5, 6, and 8; Second and subsequent courses: Day 5 only

SECONDARY OUTCOMES:
Global safety profile of SAR103168 based on treatment emergent adverse events (TEAEs), serious adverse events (SAEs), deaths, laboratory abnormalities | Treatment period up to 1 year
Preliminary evidence of anti-leukemia activity | Treatment period up to 1 year
Pharmacokinetic parameters of midazolam in the absence and the presence of SAR103168. | During second (Day-1 and Day 5) and forth course (Day 5)

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, MD, Principal Investigator — M.D. Anderson Cancer Center, Houston, Texas
Locations (3):
- United States (3):
  - Sanofi-Aventis Investigational Site Number 840003, Atlanta, Georgia
  - Sanofi-Aventis Investigational Site Number 840002, New York, New York
  - Sanofi-Aventis Investigational Site Number 840001, Houston, Texas

REFERENCES:
- [Derived] Roboz GJ, Khoury HJ, Jabbour E, Session W, Ritchie EK, Miao H, Faderl S, Zheng W, Feldman EJ, Arellano M, Morrison JG, Ravandi F. Phase I trial of SAR103168, a novel multi-kinase inhibitor, in patients with refractory/relapsed acute leukemia or high-risk myelodysplastic syndrome. Leuk Lymphoma. 2015 Feb;56(2):395-400. doi: 10.3109/10428194.2014.918970. PMID 24794806